CLINICAL TRIAL: NCT01489579
Title: Evaluation of Brief, Structured, Telephone Counseling for Tobacco Cessation as Part of a Cardiovascular Risk Reduction Service
Brief Title: Telephone Counseling for Tobacco Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CO-11-1660
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BST counseling group (Active Comparator): The patients in the Brief, structured, telephone tobacco cessation, BST, counseling group, will receive tobacco cessation counseling, intervention, by a trained CPCRS pharmacist as part of their routine CPCRS care. The counseling will not be scripted, but must contain three key components (recommendation to quit, discussion/recommendation of tobacco cessation medications, and discussion/recommendation of tobacco cessation methods/strategies (Appendix C). These are the same items measured by the National Committee for Quality Assurance (NCQA) for Healthcare Effectiveness and Data Information Set (HEDIS) reporting. A standard KPCO document will be mailed to the patients following the BST counseling containing information about available resources.
  Interventions: Behavioral: Telephone Counseling for Tobacco Cessation
- Usual care group (Placebo Comparator): Pharmacists randomized to Usual Care will continue to provide interventions/procedures they normally would according to usual care practices. These interventions include any of the following: no action, mailed information on the resources available to help aid tobacco cessation, telephone counseling, and/or assistance in getting tobacco cessation medications. Pharmacists who are randomized to Usual Care will be asked to continue their current approach for tobacco cessation recommendations
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Telephone Counseling for Tobacco Cessation — The patients in the Brief, Structured, Telephone (BST) counseling group will receive tobacco cessation counseling by a trained CPCRS pharmacist as part of their routine CPCRS care. The counseling will not be scripted, but must contain three key components (recommendation to quit, discussion/recommendation of tobacco cessation medications, and discussion/recommendation of tobacco cessation methods/strategies (Appendix C). These are the same items measured by the National Committee for Quality Assurance (NCQA) for Healthcare Effectiveness and Data Information Set (HEDIS) reporting. A standard KPCO document will be mailed to the patients following the BST counseling containing information about available resources ("Ready to quit" patient handout)
  Arms: BST counseling group
Behavioral: Usual Care — Pharmacists randomized to Usual Care will continue to provide interventions/procedures they normally would according to usual care practices. These interventions include any of the following: no action, mailed information on the resources available to help aid tobacco cessation, telephone counseling, and/or assistance in getting tobacco cessation medications. Pharmacists who are randomized to Usual Care will be asked to continue their current approach for tobacco cessation recommendations
  Arms: Usual care group

SUMMARY:
The purpose of this study is to determine whether giving more structured information to patients over the phone about quitting tobacco helps to increase the chance that they will try to quit. The results of this study will help provide direction in developing a more standard way of helping patients to quit.

Study Hypothesis:

Brief, structured, telephone tobacco cessation counseling delivered by clinical pharmacy specialists will significantly increase the percentage of self-reported tobacco cessation attempts compared to usual care among patients enrolled in a cardiovascular risk reduction program.

DETAILED DESCRIPTION:
While physician-delivered care may have the greatest impact on tobacco abstinence rates, recent data indicate that other health care providers such as nurses and pharmacists improve tobacco abstinence rates more than self-help and/or no intervention.5 Thus, pharmacists continue to expand their clinical practice areas to include smoking cessation interventions. A meta-analysis of studies involving pharmacist-delivered smoking cessation services found quit rates at 6 to12 months follow-up ranged from 14% to16%.6 The results of this meta-analysis demonstrate that pharmacists can successfully deliver tobacco-cessation interventions and the evidence strongly suggests they are effective in helping increase tobacco cessation rates. Proactive telephone counseling can be more effective at increasing tobacco abstinence rates than self-help or no intervention.5 Telephone counseling is an effective system to help increase tobacco abstinence rates for a variety of reasons. From the tobacco user's standpoint, there are no transportation inconveniences and fewer scheduling conflicts. In addition, receiving counseling in the privacy of one's own home provides treatment access to individuals who are less willing to seek out counseling. At Kaiser Permanente Colorado (KPCO), members with a history of CVD are enrolled in the Clinical Pharmacy Cardiac Risk Service (CPCRS). The CPCRS is a clinical pharmacy specialist-managed, physician-directed program which provides secondary prevention care to over 14,000 patients. Clinical care includes evaluating and treatment of major cardiovascular risk factors, including tobacco use, for members. Currently, CPCRS has no standard of care with regard to addressing tobacco use. Clinical pharmacy specialists working in CPCRS deliver tobacco cessation advice at their own discretion, through various methods. The purpose of this pilot study is to determine whether brief, structured, telephone tobacco cessation counseling delivered by a clinical pharmacy specialist increases the number of smoking cessation attempts compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria will be eligible for the study:

* Enrolled in CPCRS at the time of counseling (12/11-02/12),
* Current tobacco user as noted in KP HealthConnect as of the date of the routine CPCRS evaluation and counseling. For study purposes, tobacco use includes any use of cigarettes, pipe, cigars, snuff, and chew.
* Continuous KPCO Denver/Boulder membership during study time period

Exclusion Criteria:

* Patients who meet any of the following criteria will not be enrolled in the study:
* <18 years of age,
* Non-English speakers,
* Deceased at time of survey, and/or
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Cymbala, PharmD, BCPS, Principal Investigator — Kaiser Permanente
Locations (1):
- Clinical Pharmacy Specialist, Clinical Pharmacy Cardiac Risk Service - Kaiser Permanente of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 347 patients were identified as eligible for study participation study personnel contacted the patient by telephone approximately 2 weeks prior to her or his scheduled SOC encounter to describe the study and obtain verbal consent for enrollment. 192 were consented.
Pre-assignment Details: Seventy-two subjects did not obtain scheduled laboratory data or have contact with a clinical pharmacist during the study time period resulting in 120 subjects, 56 and 64 in the control and intervention groups, respectively, enrolled in the study.
Groups:
- Usual Care Group: Pharmacists randomized to Usual Care will continue to provide interventions/procedures according to usual care practices. Interventions include any of the following: no action, mailed information on the resources available to help aid tobacco cessation, telephone counseling, and/or assistance in getting tobacco cessation medications. Pharmacists randomized to Usual Care were asked to continue their current approach for tobacco cessation
- BST Counseling Group: The patients in the BST counseling group will receive tobacco cessation counseling by a trained CPCRS pharmacist as part of their routine CPCRS care. The counseling will not be scripted, but must contain three key components (recommendation to quit, discussion/recommendation of tobacco cessation medications, and discussion/recommendation of tobacco cessation methods/strategies (Appendix C). These are the same items measured by the National Committee for Quality Assurance (NCQA) for Healthcare Effectiveness and Data Information Set (HEDIS) reporting. A standard KPCO document will be mailed to the patients following the BST counseling containing information about available resources
Period: Overall Study
Arm/Group | Usual Care Group | BST Counseling Group
Started | 56 | 64
Completed | 47 | 57
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- BST Counseling Group: The patients in the BST counseling group will receive tobacco cessation counseling by a trained CPCRS pharmacist as part of their routine CPCRS care. The counseling will not be scripted, but must contain three key components (recommendation to quit, discussion/recommendation of tobacco cessation medications, and discussion/recommendation of tobacco cessation methods/strategies (Appendix C). These are the same items measured by the National Committee for Quality Assurance (NCQA) for Healthcare Effectiveness and Data Information Set (HEDIS) reporting. A standard KPCO document will be mailed to the patients following the BST counseling containing information about available resources ("Ready to quit" patient handout. Brief, Structured, Telephone Counseling for Tobacco Cessation as Part of a Cardiovascular Risk Reduction Service: The patients in the BST counseling group will receive tobacco cessation counseling by a trained CPCRS pharmacist as part of their routine CPCRS care. The counse
- Usual Care Group: Pharmacists randomized to Usual Care will continue to provide interventions/procedures they normally would according to usual care practices. These interventions include any of the following: no action, mailed information on the resources available to help aid tobacco cessation, telephone counseling, and/or assistance in getting tobacco cessation medications. Pharmacists who are randomized to Usual Care will be asked to continue their current approach for tobacco cessation recommendations. Usual Care: Pharmacists randomized to Usual Care will continue to provide interventions/procedures they normally would according to usual care practices. These interventions include any of the following: no action, mailed information on the resources available to help aid tobacco cessation, telephone counseling, and/or assistance in getting tobacco cessation medications. Pharmacists who are randomized to Usual Care will be asked to continue their current approach for tobacco cessation recommendatio
- Total: Total of all reporting groups
Arm/Group | BST Counseling Group | Usual Care Group | Total
Number analyzed (Participants) | 64 | 56 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (8.1) | 64.6 (9.4) | 65.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 44
  Male | 36 | 40 | 76
Region of Enrollment [Number; unit: participants]
  United States | 64 | 56 | 120

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Self-reported Tobacco Cessation Attempts Between Groups
Description: The proportion of patients in each group who report a tobacco cessation attempt during the follow-up telephone survey conducted three months following pharmacist contact
Time Frame: 3 months
Population: Reported not smoking at follow up survey
Measure: Number; unit: participants
Groups:
- BST Counseling Group: The patients in the Brief, Structured, Telephone, BST, counseling group will receive tobacco cessation counseling by a trained CPCRS pharmacist as part of their routine CPCRS care. The counseling will not be scripted, but must contain three key components (recommendation to quit, discussion/recommendation of tobacco cessation medications, and discussion/recommendation of tobacco cessation methods/strategies (Appendix C). These are the same items measured by the National Committee for Quality Assurance (NCQA) for Healthcare Effectiveness and Data Information Set (HEDIS) reporting. A standard KPCO document will be mailed to the patients following the BST counseling containing information about available resources
Arm/Group | BST Counseling Group | Usual Care Group
Number analyzed (Participants) | 57 | 47
participants | 8 | 5

2. Secondary Outcome: The Proportion of Patients in Each Group Who Participate in the Colorado Quitline (COQL) Within Three Months of Pharmacist Contact
Description: Information on COQL participation was obtained from a prevention department within KPCO that tracks these data. Report was provided to capture who from study had participated in the COQL within 3 months of pharmacist contact.
Time Frame: 3 months
Population: Three control patients reported participation in the Colorado quitline
Measure: Count of Participants; unit: Participants
Arm/Group | BST Counseling Group | Usual Care Group
Number analyzed (Participants) | 64 | 56
Participants | 0 | 3

3. Secondary Outcome: The Proportion of Patients Who Attend Any KPCO Tobacco Cessation Program(s)or Webinar(s) Within Three Months Following Contact.
Description: The proportion of patients who attend any KPCO tobacco cessation program(s)or webinar(s) within three months following contact. Classes include Stop Smoking the Basics and Freedom from Cigarettes. Webinars include Break Free and Freedom from Tobacco
Time Frame: 3 months
Population: The proportion of patients who attend any KPCO tobacco cessation program(s)or webinar(s) within three months following contact. Classes include Stop Smoking the Basics and Freedom from Cigarettes. Webinars include Break Free and Freedom from Tobacco
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care Group: The study arms were balanced on baseline characteristics except for the control arm having a higher median chronic disease score (P = 0.013) Sixteen subjects (9 and 7 in the control and intervention arms, respectively) did not complete the follow-up tele- phone survey, resulting in 104 subjects (47 and 57 in the control and intervention arm, respectively) available for the survey-based outcome analyses. Cigarettes were the predominate type of tobacco used. Fewer than half of the subjects reported ''Yes'' to baseline readiness to quit in the next 30 days. There were no statistically significant differences identified in the primary (P = 0.804) or secondary outcomes (all P > 0.05)
Arm/Group | BST Counseling Group | Usual Care Group
Number analyzed (Participants) | 64 | 56
Participants | 1 | 0

4. Secondary Outcome: The Proportion of Patients in Each Group Who Purchase Tobacco Cessation Medication Aids From KPCO Pharmacies Within Three Months Following Pharmacist Contact.
Description: The proportion of patients in each group who purchase tobacco cessation medication aids from KPCO pharmacies within three months following pharmacist contact. Medications include nicotine replacement therapy, bupropion, and varenicline
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | BST Counseling Group | Usual Care Group
Number analyzed (Participants) | 64 | 56
Participants | 7 | 11

5. Secondary Outcome: The Proportion of Patients in Each Group Who Report Tobacco Abstinence During at the Three Months Follow-up Telephone Survey
Description: The proportion of patients in each group who report tobacco abstinence during the follow-up telephone survey conducted three months following pharmacist contact
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | BST Counseling Group | Usual Care Group
Number analyzed (Participants) | 57 | 47
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: 3 month follow up
Groups:
- BST Counseling Group: The patients in the BST counseling group will receive tobacco cessation counseling by a trained CPCRS pharmacist as part of their routine CPCRS care. The counseling will not be scripted, but must contain three key components (recommendation to quit, discussion/recommendation of tobacco cessation medications, and discussion/recommendation of tobacco cessation methods/strategies (Appendix C). These are the same items measured by the National Committee for Quality Assurance (NCQA) for Healthcare Effectiveness and Data Information Set (HEDIS) reporting. A standard KPCO document will be mailed to the patients following the BST counseling containing information about available resources. AE's captured for patients who obtained lab data and had contact with clinical Pharmacist (120)
- Usual Care Group: Pharmacists randomized to Usual Care will continue to provide interventions/procedures they normally would according to usual care practices. These interventions include any of the following: no action, mailed information on the resources available to help aid tobacco cessation, telephone counseling, and/or assistance in getting tobacco cessation medications. Pharmacists who are randomized to Usual Care will be asked to continue their current approach for tobacco cessation recommendations. AE's captured for patients who obtained lab data and had contact with clinical Pharmacist (120)
Arm/Group | BST Counseling Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/56
Other Adverse Events (participants affected / at risk) | 0/64 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No